CLINICAL TRIAL: NCT03621475
Title: Pilot Study of a Novel Arm Restraint For Critically Ill Patients
Brief Title: Novel Arm Restraint in the Intensive Care Unit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Healthy Design, LLC (Unknown)
Responsible Party: Principal Investigator, Renee Stapleton, Associate Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 18-0353-01
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel restraint first, then traditional restraint (Experimental): Participants will be randomized to wear the novel arm restraint bilaterally for 4 hours on study day #1, followed by traditional soft bilateral wrist restraints for 4 hours. Then, on study day #2, they will wear both kinds of restraints in the opposite order.
  Interventions: Device: Novel restraint
- Traditional restraint first, then novel restraint (Experimental): Participants will be randomized to wear traditional soft bilateral wrist restraints for 4 hours on study day #1, followed by the novel arm restraint bilaterally for 4 hours. Then, on study day #2, they will wear both kinds of restraints in the opposite order.
  Interventions: Device: Novel restraint

INTERVENTIONS:
Device: Novel restraint — Use of a novel arm restraint

SUMMARY:
The goal of this pilot is to evaluate a novel restraint device in 8 older mechanically ventilated patients to demonstrate that 1) the revised novel restraint prototype is safe and 2) a future randomized controlled trial (RCT) is feasible.

DETAILED DESCRIPTION:
The goal of this Fast-Track Small Business Technology Transfer (STTR) project is to optimize and test a novel arm restraint in older critically ill mechanically ventilated patients that may increase mobility; reduce agitation, use of sedative medications, and delirium; and exhibit high satisfaction and acceptability among hospital staff, family members, and patients. Older mechanically ventilated patients are often immobilized with wrist restraints to prevent self-extubation and are sedated to reduce agitation caused by their restraints and endotracheal (breathing) tube. This sedation and immobility lead to complications, including delirium and muscle weakness, that are independently associated with long term cognitive impairment, reduced physical functioning, and mortality. Specifically, the incidence and duration of delirium in the ICU are strongly and independently associated with long-term cognitive impairment that is similar to Alzheimer's Disease and Related Dementias.

Healthy Design has developed a novel restraint device that allows arm mobility but prohibits hands from reaching oral/nasal endotracheal and feeding tubes or intravenous lines. Because it permits mobility, the novel restraint may reduce agitation and the need for sedatives. The objectives of this pilot study are to evaluate the novel restraint in 8 older mechanically ventilated patients to demonstrate that 1) the revised novel restraint prototype is safe and 2) a future RCT is feasible.

ELIGIBILITY:
Inclusion Criteria:

1. >65 years old
2. Physician order for use of bilateral wrist restraints
3. Requiring mechanical ventilation with actual or expected total duration of >48 hours
4. Expected ICU stay >3 days after enrollment (to permit adequate exposure to proposed intervention)
5. Not deeply sedated (Richmond Agitation Sedation Scale [RASS] score > -2)

Exclusion Criteria:

1. Upper extremity impairments that prevent use of novel restraint device (e.g. amputation, arm injury)
2. Limited mobility of either upper extremity prior to admission (e.g. frozen shoulder, severe arthritis)
3. Pre-existing primary systemic neuromuscular disease (e.g. Guillain-Barre)
4. Neuromuscular blocker infusion (eligible once infusion discontinued if other inclusion criteria met)
5. Pre-existing severe cognitive impairment or language barrier prohibiting outcome assessment
6. Expected death or withdrawal of life-sustaining treatments within 6 days from enrollment
7. Incarcerated
8. Severe skin breakdown on either upper extremity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In two academic ICUs within the same medical center, non-comatose, mechanically ventilated adults >25 years old who required restraints and had an expected ICU stay of at least 2 days were evaluated for eligibility. The recruitment period was 10/2/2018 -- 4/8/2019.
Groups:
- Novel Restraint First, Then Traditional Restraint: Participants were randomized to wear the novel arm restraint bilaterally for 4 hours on study day #1, followed by traditional soft bilateral wrist restraints for 4 hours. Then, on study day #2, they wore both kinds of restraints in the opposite order.
  Novel restraint: Use of a novel arm restraint
- Traditional Restraint First, Then Novel Restraint: Participants were randomized to wear traditional soft bilateral wrist restraints for 4 hours on study day #1, followed by the novel arm restraint bilaterally for 4 hours. Then, on study day #2, they wore both kinds of restraints in the opposite order.
  Novel restraint: Use of a novel arm restraint
Period: Overall Study
Arm/Group | Novel Restraint First, Then Traditional Restraint | Traditional Restraint First, Then Novel Restraint
Started | 4 | 4
Completed | 4 | 3
Not Completed | 0 | 1
Not completed — No longer required restraints at initiation | 0 | 1

BASELINE CHARACTERISTICS:
Population: participants
Groups:
- Novel Restraint First, Then Traditional Restraint: Crossover design in which participants were randomized to wear the novel arm restraint bilaterally for 4 hours on study day #1, followed by traditional soft bilateral wrist restraints for 4 hours. Then, on study day #2, they wore both kinds of restraints in the opposite order.
  Novel restraint: Use of a novel arm restraint
- Traditional Restraint First, Then Novel Restraint: Crossover design in which participants were randomized to wear the traditional arm restraint bilaterally for 4 hours on study day #1, followed by novel soft bilateral wrist restraints for 4 hours. Then, on study day #2, they wore both kinds of restraints in the opposite order.
  Novel restraint: Use of a novel arm restraint
- Total: Total of all reporting groups
Arm/Group | Novel Restraint First, Then Traditional Restraint | Traditional Restraint First, Then Novel Restraint | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Customized [Median (Full Range); unit: years] | 65.5 [49 to 73] | 64 [55 to 70] | 65 [49 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Severe Adverse Events [Safety]
Description: Safety will be measured by the number (i.e. < 1 in 5 participants had a treatment emergent safety event per their on study time) across all of the following measures listed below. Incidence does not have to be per person-year; in this case it is incidence of safety adverse event during the study period.
Time Frame: Through study day 2
Measure: Number; unit: number of safety events
Groups:
- Novel Restraint: Crossover design of novel and traditional hospital restraints. 7 participants wore the novel restraint.
- Traditional Restraint: Crossover design of novel and traditional hospital restraints. 6 participants wore the traditional restraint.
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
number of safety events | 0 | 0

2. Primary Outcome: Number of Clinician or Patient Lacerations
Description: Grade 2b or higher skin laceration (per Skin Tear Audit Research [STAR] Skin Tear Classification System) in patient or clinician from any sharp edges of device. The STAR grading system ranges from grade 1a at best to 3 at worst. Each laceration is given an individual score based on appearance.
Time Frame: Through study day 2
Measure: Number; unit: number of clinician/patient lacerations
Groups:
- Novel Restraint: Crossover design of both novel and traditional restraint devices. 7 participants wore novel restraint.
- Traditional Restraint: Crossover design of both novel and traditional restraint devices. 6 participants wore traditional restraint.
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
number of clinician/patient lacerations | 0 | 0

3. Primary Outcome: Number of Pressure Ulcers From Device
Description: Development of pressure ulcer from device of Stage 3 or greater per 2016 National Pressure Ulcer Advisory Panel Pressure Injury Stages. This staging system provides an individual score to each pressure ulcer based on appearance from stage 1 (best) to stage 4 (worst)
Time Frame: Through study day 2
Measure: Number; unit: number of pressure ulcers
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
number of pressure ulcers | 0 | 0

4. Primary Outcome: Number of Self-removals of Novel Restraint
Description: Self-removal of novel restraint
Time Frame: Through study day 2
Measure: Number; unit: number of restraint removals
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
number of restraint removals | 0 | 0

5. Primary Outcome: Number of Damaging Events to Hospital Bed Rendering it Non-functional
Description: Any damage to hospital bed from restraint device rendering it non-functional
Time Frame: Through study day 2
Measure: Number; unit: number of damage events to bed incidents
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
number of damage events to bed incidents | 0 | 0

6. Primary Outcome: Number of Damaging Events to ICU Equipment
Description: Any damage to ICU equipment (e.g. ventilator) rendering it non-functional
Time Frame: Through study day 2
Measure: Number; unit: number of damage events to ICU equipment
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
number of damage events to ICU equipment | 0 | 0

7. Secondary Outcome: Number of Self-extubations
Description: Will record instances where participants remove own endotracheal tube
Time Frame: Through study day 2
Measure: Number; unit: number of self-extubations
Groups:
- Traditional Restraint First, Then Novel Restraint: Crossover design of both novel and traditional restraint devices. 6 participants wore traditional restraint.
Arm/Group | Novel Restraint | Traditional Restraint First, Then Novel Restraint
Number analyzed (Participants) | 7 | 6
number of self-extubations | 0 | 0

8. Secondary Outcome: Number of Movements of Upper Extremities
Description: Actigraphy counts of upper extremities as measured by Philliips actigraph, a device that records individual movements
Time Frame: Continuously through study day 2
Population: Enrolled subjects who wore the restraint/restraint alternative devices
Measure: Number; unit: number of movement events
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
number of movement events | 27,509 | 24,686

9. Secondary Outcome: Richmond Agitation Sedation Score [RASS]
Description: Agitation measured by the median of Richmond agitation sedation score [RASS] collected longitudinally every hour while wearing restraints. This score measures sedation and agitation from a scale of -5 (most sedated) to +4 (most agitated)
Time Frame: Median of multiple RASS scores collected over first 2 days of study period
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Novel Restraint | Traditional Restraint
Number analyzed (Participants) | 7 | 6
score on a scale | -1.5 [-2 to 0] | -1 [-2 to -0.5]

10. Secondary Outcome: Satisfaction With Novel Device as Assessed by the Quebec User Evaluation of Satisfaction With Assistive Technology (QUEST) Satisfaction Score
Description: Satisfaction with the novel restraint device will be measured with the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) satisfaction tool. This 12-item questionnaire is scored from 1 (lowest satisfaction) to 5 (highest satisfaction).
Time Frame: Study day 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Patient Proxies, Physicians and Nurses: Proxies of enrolled patients (family members who were present at the bedside), physicians and nurses who were on the care teams for enrolled patients and were present at the bedside
Arm/Group | Patient Proxies, Physicians and Nurses
Number analyzed (Participants) | 10
score on a scale | 3.5 [2.5 to 4.25]

11. Secondary Outcome: Delerium Score
Description: We intended to measure delirium score as accessed by the CAM-ICU. However, during the study we were unable to measure it because it was too often incorrectly charted by nursing. We therefore have nothing to report for this planned outcome.
Time Frame: 6-day study period
Population: We intended to measure delirium score as accessed by the CAM-ICU. However, during the study we were unable to measure it because it was too often incorrectly charted by nursing. We therefore have nothing to report for this planned outcome.
Arm/Group | Novel Restraint First, Then Traditional Restraint | Traditional Restraint First, Then Novel Restraint
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Enrolling Adequate Numbers of Patients
Description: Number of participants enrolled in the study
Time Frame: 6-day study period
Population: participants enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Restraint First, Then Traditional Restraint | Traditional Restraint First, Then Novel Restraint
Number analyzed (Participants) | 4 | 4
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 2 days while the participants were enrolled in the study and required physical restraint as determined by the clinical team.
Groups:
- Novel Restraint; Traditional Restraint: Per intervention
Arm/Group | Novel Restraint | Traditional Restraint
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT03621475/Prot_SAP_000.pdf